CLINICAL TRIAL: NCT00712504
Title: A Phase 1 Safety And Pharmacokinetic Study Of SU011248 In Combination With Docetaxel In Patients With Advanced Solid Tumors
Brief Title: Study Of SU011248 In Combination With Docetaxel In Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181035
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Advanced Solid Tumors; Non Small Cell Lung Cancer
Keywords: advanced solid tumors, non small cell lung cancer, pulmonary neoplasms, sunitinib (SUTENT), docetaxel (Taxotere), Angiogenesis Inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Sunitinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SU011248 in combination with docetaxel
  Interventions: Drug: sunitinib; Drug: docetaxel

INTERVENTIONS:
Drug: sunitinib — 25, 37.5 and 50 mg/day, oral, administered on an outpatient basis in two different dosing regimens: schedule 2/1 (2 weeks on, 1 week off) and schedule 4/2 (4 weeks on, 2 weeks off)
Drug: docetaxel — 60, 75, and 100 mg/m2 docetaxel administered every 21 days as a 1-hr IV infusion

SUMMARY:
This study is determining the maximum tolerated dose and safety of SU011248 (sunitinib malate, SUTENT) in combination with docetaxel (Taxotere). Several dosing regimens will be tested in patients with advanced solid tumors, including non small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

Advanced solid tumor malignancy ECOG 0 or 1

Exclusion Criteria:

Prior treatment with with high-dose chemotherapy requiring stem cell rescue Prior irradiation to ≥25% of the bone marrow (e.g. whole pelvis=25%) Patients with centrally located lung lesions unless recently treated with radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity, timing, seriousness, and relatedness of adverse events and laboratory abnormalities | November 2007

SECONDARY OUTCOMES:
Pharmacokinetic parameters of SU011248 (and its active metabolite, SU012662), and docetaxel. | November 2007
Objective disease response | November 2007

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Madison, Wisconsin